CLINICAL TRIAL: NCT03080636
Title: Sex and Exercise-mode Differences in Post Exercise Blood Pressure and Heart Rate Variability Responses During Workday
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Igor Moraes Mariano, Principal Investigator, Federal University of Uberlandia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CAAE: 28174814.9.0000.5152
Record Dates: First submitted 2017-03-07; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Hemodynamic; Exercise
Keywords: Post-exercise hypotension; Aerobic Exercise; Resistance Exercise; Autonomic Stress; Heart Rate Variability; Sex difference
MeSH Terms: conditions — Motor Activity; Post-Exercise Hypotension | interventions — Exercise; Resistance Training

STUDY DESIGN:
Intervention Model Description: 20 healthy adults, public servants (9W and 11M), randomly underwent three experimental sessions in early morning prior to their work routine: a circuit resistance session at 40% of 1RM, a treadmill exercise session at 60-70% of heart rate reserve and a resting control session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Men (Experimental): 11 men randomly underwent three experimental sessions in early morning prior to their work routine.
  Interventions: Other: Aerobic exercise; Other: Resistance exercise; Other: Control session
- Women (Experimental): 9 women randomly underwent three experimental sessions in early morning prior to their work routine.
  Interventions: Other: Aerobic exercise; Other: Resistance exercise; Other: Control session

INTERVENTIONS:
Other: Aerobic exercise — 30 minutes of treadmill exercise at 60-70% of heart rate reserve
Other: Resistance exercise — 30 minutes of circuit resistance session at 40% of 1 maximun repetition test
Other: Control session — 30 minutes seated resting

SUMMARY:
The present study compared the acute effects of Sex and exercise mode on subsequent blood pressure (BP) and heart rate variability (HRV) responses during daily work in healthy adults. All subjects did 3 sessions: aerobic exercise on a treadmill, resistance exercise at the gym and a seated control session.

DETAILED DESCRIPTION:
Resting blood pressure and heart rate variability are simple and non-invasive methods to evaluate cardiovascular risk after different exercise sessions. Thus, exercise can reduce these risk factors in the short and long term, but these responses can be different between sex in different exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

* Able to practice aerobic and resistance exercise at moderate intensity;
* Men and women;
* Normotensive, pre-hypertensive or hypertensive stage 1.

Exclusion Criteria:

* Renal pathologies;
* Using beta blockers;
* History of stroke or acute myocardial infarction;
* Smokers.

Ages: 28 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-12-24 (Actual); Study Completion 2015-02-20 (Actual)

PRIMARY OUTCOMES:
Resting blood pressure | Change from baseline Systolic and Diastolic Blood Pressure to 15, 30, 45, 60, 210, 360 and 540 minutes after exercise/control session
  During all sessions, systolic (SBP) and diastolic blood pressure (DBP) were triplicate measured by an automatic blood pressure analyzer after rest in seated position.
Heart Rate Variability | Change from baseline Heart Rate Variability components to 15, 30, 45 and 60 minutes after exercise/control session
  The HR was recorded by a heart rate monitor (sampling frequency = 1000Hz) in a beat-by-beat basis. HR was registered in a seat position during 15 minutes for each measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Guilherme Morais Puga, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gomes Anunciacao P, Doederlein Polito M. A review on post-exercise hypotension in hypertensive individuals. Arq Bras Cardiol. 2011 May;96(5):e100-109. Epub 2011 Mar 4. English, Portuguese, Spanish. PMID 21359479
- [Background] Halliwill JR, Buck TM, Lacewell AN, Romero SA. Postexercise hypotension and sustained postexercise vasodilatation: what happens after we exercise? Exp Physiol. 2013 Jan;98(1):7-18. doi: 10.1113/expphysiol.2011.058065. Epub 2012 Aug 7. PMID 22872658
- [Background] Queiroz AC, Rezk CC, Teixeira L, Tinucci T, Mion D, Forjaz CL. Gender influence on post-resistance exercise hypotension and hemodynamics. Int J Sports Med. 2013 Nov;34(11):939-44. doi: 10.1055/s-0033-1337948. Epub 2013 Apr 19. PMID 23606339
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Cote AT, Bredin SS, Phillips AA, Koehle MS, Warburton DE. Greater autonomic modulation during post-exercise hypotension following high-intensity interval exercise in endurance-trained men and women. Eur J Appl Physiol. 2015 Jan;115(1):81-9. doi: 10.1007/s00421-014-2996-5. Epub 2014 Sep 11. PMID 25208772